CLINICAL TRIAL: NCT00742027
Title: A Phase II Study of Oral Panobinostat in Adult Patients With Relapsed/Refractory Classical Hodgkins Lymphoma After High-dose Chemotherapy With Autologous Stem Cell Transplant
Brief Title: Phase II Study of Oral Panobinostat in Adult Participants With Relapsed/Refractory Classical Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589E2214; 2008-003016-35 (EudraCT Number)
Record Dates: First submitted 2008-08-25; First posted 2008-08-27 (Estimated); Results first posted 2021-06-03 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Classical Hodgkin's Lymphoma
Keywords: Classical Hodgkin Lymphoma; Classical Hodgkin's Lymphoma; Hodgkin Lymphoma; Hodgkin's Lymphoma; Nodular sclerosing; Mixed-cellularity; Lymphocyte-rich; Lymphocyte depleted; HL; Classical HL; Refractory Hodgkin's Lymphoma; Refractory Hodgkin Lymphoma; Refractory HL
MeSH Terms: conditions — Hodgkin Disease | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Panobinostat (Experimental): Participants received panobinostat 40 mg, capsules, orally, thrice every week (i.e. days 1, 3 and 5), in each cycle of 21 days until unacceptable toxicity, disease progression, start of new anti-cancer therapy or withdrawal of consent (up to approximately 48 months).
  Interventions: Drug: Panobinostat

INTERVENTIONS:
Drug: Panobinostat — Panobinostat hard gelatin capsules.
  Other Names: LBH589; LBH

SUMMARY:
This study evaluated the efficacy of oral panobinostat in participants with refractory/relapsed classical Hodgkins lymphoma (HL) who have received prior treatment with high dose chemotherapy and autologous stem cell transplant. Safety of panobinostat also was assessed. Other markers that may correlate with efficacy or safety were explored.

ELIGIBILITY:
Inclusion Criteria:

1. Participant age is ≥ 18 years.
2. Participant has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
3. Participant has a history of classical Hodgkin's Lymphoma (HL) (i.e. Nodular sclerosing, Mixed-cellularity, Lymphocyte-rich, Lymphocyte depleted).
4. Participant has progressive disease after receiving high dose chemotherapy with autologous hematopoietic stem cell transplant (AHSCT).

   Note: If last therapy was ≥ 18 months ago, then biopsy should be performed to confirm diagnosis.

   Note: Participant should have received ≤ 5 prior systemic treatment regimens (See Post-text supplement 2 for definitions and examples).

   Note: Participant will be allowed on study who have also received an allogeneic hematopoietic stem cell transplant, however this therapy alone is not sufficient for inclusion into this study.
5. Participant has at least one site of measurable nodal disease at baseline ≥ 2.0 centimeter (cm) in the longest transverse diameter and clearly measurable in at least two perpendicular dimensions, as determined by computed tomography (CT) scan (magnetic resonance imaging [MRI] is allowed only if CT scan can not be performed).

   Note: Participant with bone marrow involvement are eligible, but this criteria alone should not be used for disease measurement.
6. Participant has the following laboratory values (labs may be repeated, if needed, to obtain acceptable values before screen fail):

   * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/liter (L) [International System of Units {SI} units 1.5 x 10^9/L].
   * Platelet count ≥ 75 x 10^9/L.
   * Serum potassium, magnesium, phosphorus, sodium, total calcium (corrected for serum albumin) or ionized calcium within normal limits (WNL) for the institution.

   Note: Potassium, calcium, magnesium, sodium, and/or phosphorus supplements may be given to correct values that are < lower limits of normal (LLN). Post-correction values must not be deemed to be a clinically significant abnormality prior to participant being dosed.
   * Serum creatinine ≤ 1.5 x upper limits of normal (ULN).
   * Serum bilirubin ≤ 1.5 x ULN (or ≤ 3.0 x ULN, if participant has Gilbert syndrome).
   * Aspartate transaminase (AST)/ serum glutamic oxaloacetic transaminase (SGOT) and/or alanine transaminase (ALT)/ serum glutamic pyruvic transaminase (SGPT) ≤ 2.5 x ULN or ≤ 5.0 x ULN if the transaminase elevation is due to disease involvement.
7. Clinically euthyroid. Note: Participants are permitted to receive thyroid hormone supplements to treat underlying hypothyroidism.
8. Written informed consent was obtained from the participant prior to any study-specific screening procedures.
9. Participant has the ability to swallow capsules or tablets.

Exclusion Criteria:

1. Participant has a history of prior treatment with a deacetylase (DAC) inhibitor including panobinostat.
2. Participant will need valproic acid for any medical condition during the study or within 5 days prior to the first panobinostat treatment.
3. Participant has been treated with monoclonal antibody therapy (e.g., rituximab or anti CD-30 antibody, etc.) within 4 weeks of start of study treatment.
4. Participant has received chemotherapy or any investigational drug or undergone major surgery ≤ 2 weeks prior to starting study drug or whose side effects of such therapy have not resolved to ≤ grade 1.
5. Participant has been treated with > 5 prior systemic lines of treatment (see Post-text supplement 2 for definitions and examples).
6. Participant has received prior radiation therapy ≤ 4 weeks or limited field radiotherapy ≤ 2 weeks prior to start of study treatment or whose side effects of such therapy have not resolved to ≤ grade 1.
7. Participant is using any anti-cancer therapy concomitantly.
8. Participant treated with allogeneic hematopoietic stem cell transplant who is currently on or has received immunosuppressive therapy within 90 days prior to start of screening and/or have ≥ Grade 2 graft versus host disease (GvHD).
9. Participant has a history of another primary malignancy ≤ 3 years before study entry, with the exception of non-melanoma skin cancer, and carcinoma in situ of uterine cervix.
10. Participant has a history of central nervous system (CNS) involvement with lymphoma.
11. Participant has impaired cardiac function including any of the following:

    * Complete left bundle branch block or use of a permanent cardiac pacemaker, congenital long QT syndrome, history or presence of ventricular tachyarrhythmias, clinically significant resting bradycardia (<50 beats per minute [bpm]), QT interval (QTcF) > 450 milliseconds (msec) on screening electrocardiography (ECG), or right bundle branch block + left anterior hemiblock (bifascicular block).
    * Presence of atrial fibrillation (ventricular heart rate >100 bpm).
    * Previous history angina pectoris or acute myocardial infarction (MI) within 6 months.
    * Congestive heart failure (New York Heart Association functional classification III-IV) or baseline multigated acquisition (MUGA)/Echo shows left ventricular ejection fraction (LVEF) < 45%.
12. Participant has any other clinically significant heart disease (e.g., uncontrolled hypertension).
13. Participant has an impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of panobinostat (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, obstruction, or stomach and/or small bowel resection).
14. Participant has unresolved diarrhea ≥ grade 2.
15. Participant has any other concurrent severe and/or uncontrolled medical condition(s) (e.g., uncontrolled diabetes mellitus, active or uncontrolled infection, chronic obstructive or chronic restrictive pulmonary disease including dyspnoea at rest from any cause) that could cause unacceptable safety risks or compromise compliance with the protocol.
16. Participant has a known history of human immunodeficiency virus (HIV) seropositivity (screening HIV testing is not required).
17. Participant is using medications that have a relative risk of prolonging the QT interval or of inducing Torsade de Pointes, where such treatment cannot be discontinued or switched to a different medication prior to starting study drug.
18. Participant is a woman who is pregnant or breast feeding, or a women of childbearing potential (WOCBP) not willing to use a double method of contraception during the study through 3 months after the end of treatment. One of these methods of contraception must be a barrier method. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months). WOCBP must have a negative serum pregnancy test at baseline.
19. Male participant whose sexual partner(s) are WOCBP who are not willing to use a double method of contraception, one of which includes a condom, during the study and for 3 months after the end of treatment.

    Participants with any of the following contraindications to positron emission tomography (PET) are excluded from the [18F]- fludeoxyglucose (FDG) PET study (only applicable for centers participating in the PET study):
20. Fasting blood glucose above 200 milligrams per deciliter (mg/dL), at time of PET scan.
21. Inability to lay down for 60 minutes or has a history of claustrophobia.
22. Participant not at a participating center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2008-09-16 (Actual); Primary Completion 2013-08-12 (Actual); Study Completion 2013-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (45):
- United States (13):
  - City of Hope National Medical Center Dept.ofCityofHopeMedicalCtr(2), Duarte, California
  - Emory University School of Medicine/Winship Cancer Institute Dept. of Hematology (2), Atlanta, Georgia
  - Georgia Regents University Cancer Clinical Research Unit, Augusta, Georgia
  - Rush University Medical Center Divisionof Hem/Onc Research(2), Chicago, Illinois
  - VA Maryland Health Care Dept.of GreenbaumCancerCent(5), Baltimore, Maryland
  - Dana Farber Cancer Institute Hematology / Oncology, Boston, Massachusetts
  - Karmanos Cancer Institute Div.of Hematology/Oncology, Detroit, Michigan
  - Mayo Clinic - Rochester Hematology, Rochester, Minnesota
  - University of Pennsylvania Medical Center Dept of UPenn Med Ctr (3), Philadelphia, Pennsylvania
  - University of Texas/MD Anderson Cancer Center Dept.ofMDAndersonCancerCtr(3), Houston, Texas
  - The Methodist Hospital Cell & Gene Therapy Clinic, Houston, Texas
  - Cancer Therapy & Research Center / UT Health Science Center InstituteForDrugDevelopment(5), San Antonio, Texas
  - West Virginia University/ Mary Babb Randolph Cancer Center, Morgantown, West Virginia
- Australia (2):
  - Novartis Investigative Site, Herston, Queensland
  - Novartis Investigative Site, Malvern, Victoria
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, Leuven
- Brazil (3):
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- France (6):
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Villejuif
- Germany (3):
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Göttingen
- Israel (3):
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Ramat Gan
- Italy (5):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Udine, UD
- Novartis Investigative Site, Kuala Selangor, Malaysia
- Novartis Investigative Site, Auckland, New Zealand
- Novartis Investigative Site, Singapore, Singapore
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- United Kingdom (2):
  - Novartis Investigative Site, Withington, Greater Manchester
  - Novartis Investigative Site, Southampton

REFERENCES:
- [Derived] Chari A, Cho HJ, Dhadwal A, Morgan G, La L, Zarychta K, Catamero D, Florendo E, Stevens N, Verina D, Chan E, Leshchenko V, Lagana A, Perumal D, Mei AH, Tung K, Fukui J, Jagannath S, Parekh S. A phase 2 study of panobinostat with lenalidomide and weekly dexamethasone in myeloma. Blood Adv. 2017 Aug 21;1(19):1575-1583. doi: 10.1182/bloodadvances.2017007427. eCollection 2017 Aug 22. PMID 29296798
- [Derived] Harrison SJ, Hsu AK, Neeson P, Younes A, Sureda A, Engert A, Prince HM, Li M, Savage P, Bugarini R, Williams D, Squier M, Ritchie DS. Early thymus and activation-regulated chemokine (TARC) reduction and response following panobinostat treatment in patients with relapsed/refractory Hodgkin lymphoma following autologous stem cell transplant. Leuk Lymphoma. 2014 May;55(5):1053-60. doi: 10.3109/10428194.2013.820287. Epub 2013 Aug 5. PMID 23822537

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 45 sites in 13 countries from 16 September 2008 to 12 August 2013.
Pre-assignment Details: A total of 102 participants were to be enrolled and treated in the study. However, 129 participants got enrolled and analyzed, out of which no participant completed the study.
Period: Overall Study
Arm/Group | Panobinostat
Started | 129
Completed (Deaths reported included deaths that occurred more than 28 days after treatment discontinuation.) | 0
Not Completed | 129
Not completed — Disease Progression | 76
Not completed — New Cancer Therapy | 19
Not completed — Withdrawal by Subject | 18
Not completed — Death | 7
Not completed — Lost to Follow-up | 4
Not completed — Follow up Phase Completed As Per Protocol | 2
Not completed — Missing | 2
Not completed — Administrative Problems | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who received at least one dose of study drug.
Arm/Group | Panobinostat
Number analyzed (Participants) | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (12.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 66

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) as Assessed by the Investigator Based on Cheson Response Criteria
Description: ORR was number of participants with best overall disease response of complete response(CR)/partial response(PR).Best overall disease response was best disease response recorded from start of treatment until disease progression/recurrence.CR=complete normalization of all index nodal,extranodal lesions,complete disappearance of all extranodal lesions.PR=50% decrease in SPD for up to 6 identified dominant lesions (splenic,hepatic nodules) from baseline.Stable=neither sufficient shrinkage to qualify for PR nor sufficient increase for progressive disease (PD), reference smallest sum diameters while on study.Progression=50% increase in sum of longest diameter of all target lesions,from smallest sum of longest diameter of all target lesions recorded at or after baseline/a new lesion/progression of non-target lesions.Unknown is progression not documented,one/more of index lesions not assessed or have been assessed using a different method than baseline at the time of radiologic evaluation.
Time Frame: From the start of the treatment of last participant up to 32 weeks
Population: Full analysis set (FAS) included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat
Number analyzed (Participants) | 129
Participants
  Complete Response | 5
  Partial Response | 30
  Stable Disease | 71
  Progressive Disease | 14
  Unknown | 9

2. Secondary Outcome: Response Rate Based on Central Review of Computed Tomography (CT) Scan/Magnetic Resonance Imaging (MRI)
Description: Best overall radiological response (CT/MRI) was recorded from start of treatment until progression/ recurrence. CR=complete normalization of all index nodal,extranodal lesions,complete disappearance of all extranodal lesions.PR=50% decrease in SPD for up to 6 identified dominant lesions (splenic,hepatic nodules) from baseline.Stable=neither sufficient shrinkage to qualify for PR nor sufficient increase for progressive disease (PD), reference smallest sum diameters while on study.Progression=50% increase in sum of longest diameter of all target lesions,from smallest sum of longest diameter of all target lesions recorded at or after baseline/a new lesion/progression of non-target lesions.Unknown is progression not documented,one/more of index lesions not assessed or have been assessed using a different method than baseline at the time of radiologic evaluation.
Time Frame: From start of treatment until progression/recurrence or start of a new cancer therapy (up to approximately 5 years)
Population: FAS included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Panobinostat
Number analyzed (Participants) | 129
percentage of participants
  Complete Response | 0.8
  Partial Response | 20.9
  Stable Disease | 56.6
  Progressive Disease | 15.5
  Unknown | 6.2

3. Secondary Outcome: Time To Overall Disease Response in Responders
Description: Time to overall disease response (CR or PR) was defined as the time from the date of randomization/start of treatment to the date of first documented disease response (PR or CR). Per Cheson response criteria, CR= is a complete normalization of all index nodal and extranodal lesions and complete disappearance of all extranodal lesions. PR= is a 50% decrease in the SPD for up to 6 identified dominant lesions, including splenic and hepatic nodules from baseline. Participants were considered responders if they had a partial or complete response to a treatment while in the study as per Investigator's assessment.
Time Frame: From the start of treatment up to approximately 5 years
Population: FAS included all participants who received at least one dose of study drug. Participants who were responders among those who were had relapsed/refractory classical Hodgkin's lymphoma were evaluated for this outcome measure. Time to overall disease response was calculated by Kaplan-Meier estimation.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Panobinostat
Number analyzed (Participants) | 35
weeks | 9.9 [6.0 to 12.1]

4. Secondary Outcome: Duration of Overall Disease Response
Description: Duration of overall response (CR or PR) was defined as the time from the date of first documented disease response (CR or PR) to the date of first documented progression or death due to lymphoma. Per Cheson response criteria, CR= is a complete normalization of all index nodal and extranodal lesions and complete disappearance of all extranodal lesions. PR= is a 50% decrease in the SPD for up to 6 identified dominant lesions, including splenic and hepatic nodules from baseline. Participants were considered responders if they had a partial or complete response to a treatment while in the study.
Time Frame: From the start of treatment up to approximately 5 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Panobinostat
Number analyzed (Participants) | 35
weeks | 30.1 [17.4 to 35.9]

5. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival (PFS) was defined as the time from the date of randomization/start of treatment to the date of event defined as the first documented progression or death due to any cause. If a participant has not had an event, progression-free survival was censored at the date of the last adequate assessment.
Time Frame: From the start of treatment up to approximately 5 years
Population: FAS included all participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panobinostat
Number analyzed (Participants) | 129
months | 6.1 [5.4 to 8.3]

6. Secondary Outcome: The Overall Survival (OS)
Description: OS was the duration from date of randomization to date of death from any cause. If a participant has not had an event, overall survival was censored at the date of the last adequate assessment.
Time Frame: Baseline to date of death from any cause (up to approximately 5 years)
Population: FAS included all participants who received at least one dose of study drug.
Measure: Median (Full Range); unit: months
Arm/Group | Panobinostat
Number analyzed (Participants) | 129
months | 34.9 [0.7 to 53]

7. Secondary Outcome: Percentage of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), And Deaths as a Measure of Safety and Tolerability of Panobinostat
Description: An AE is the appearance of (or worsening of any pre-existing) undesirable sign(s), symptom(s), or medical condition(s) occurring after signing the informed consent even if the event is not considered to be related to the study drug(s). SAEs are AEs leading to death, are life-threatening, require hospitalizations or prolongation of hospitalizations, represent an innate malformation or a congenital abnormality.
Time Frame: Up to approximately 5 years
Population: Safety set population included all participants who received at least one dose of study drug and had at least one valid post-baseline safety assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Panobinostat
Number analyzed (Participants) | 129
percentage of participants
  AEs | 100
  SAEs | 39.5
  Deaths | 45.0

8. Secondary Outcome: Maximum Observed Concentration (Cmax) of Panobinostat
Time Frame: Cycle 1, Day 1: Pre-dose, 0.25, 1, 3, 5, 7, 24, and 28 hours post-dose
Population: Pharmacokinetic set (PK) included all participants who have received at least one dose of panobinostat and had sufficient and evaluable blood samples for the Day 1 PK profile.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Panobinostat
Number analyzed (Participants) | 13
nanograms per milliliter (ng/mL) | 41.88 (22.165)

9. Secondary Outcome: The Time to Reach Maximum Plasma Concentration (Tmax) of Panobinostat
Time Frame: Cycle 1, Day 1: Pre-dose, 0.25, 1, 3, 5, 7, 24, and 28 hours post-dose
Population: PK population included all participants who have received at least one dose of panobinostat and had sufficient and evaluable blood samples for the Day 1 PK profile.
Measure: Median (Full Range); unit: hours
Arm/Group | Panobinostat
Number analyzed (Participants) | 13
hours | 1.1 [0.30 to 6.10]

10. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to 28 Hours (AUC0-28) for Panobinostat
Time Frame: Cycle 1, Day 1: Pre-dose, 0.25, 1, 3, 5, 7, 24, and 28 hours post-dose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hour*nanograms per milliliter (h.ng/mL)
Arm/Group | Panobinostat
Number analyzed (Participants) | 13
hour*nanograms per milliliter (h.ng/mL) | 233.38 (112.138)

11. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-∞) for Panobinostat
Time Frame: Cycle 1, Day 1: Pre-dose, 0.25, 1, 3, 5, 7, 24, and 28 hours post-dose
Population: PK population included all participants who have received at least one dose of panobinostat and had sufficient and evaluable blood samples for the Day 1 PK profile. Overall number analyzed is the number of participants with data available for this analyses.
Measure: Mean (Standard Deviation); unit: h.ng/mL
Arm/Group | Panobinostat
Number analyzed (Participants) | 11
h.ng/mL | 239.36 (104.263)

ADVERSE EVENTS:
Time Frame: Up to approximately 5 years
Description: Safety set population included all participants who received at least one dose of study drug and had at least one valid post-baseline safety assessment.
Arm/Group | Panobinostat
Serious Adverse Events (participants affected / at risk) | 51/129
Other Adverse Events (participants affected / at risk) | 129/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panobinostat (N=129)
Anaemia (Blood and lymphatic system disorders) | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Haemorrhagic disorder (Blood and lymphatic system disorders) | 1
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 12
Atrial fibrillation (Cardiac disorders) | 3
Pericardial effusion (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Ventricular hypokinesia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Multi-organ failure (General disorders) | 1
Pyrexia (General disorders) | 2
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Appendicitis (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Dengue fever (Infections and infestations) | 1
Device related infection (Infections and infestations) | 2
Device related sepsis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 2
Necrotising ulcerative gingivostomatitis (Infections and infestations) | 1
Neutropenic sepsis (Infections and infestations) | 1
Oropharyngeal candidiasis (Infections and infestations) | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Pneumonia pneumococcal (Infections and infestations) | 1
Sepsis (Infections and infestations) | 4
Septic shock (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Cachexia (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Cervicitis human papilloma virus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Intracranial venous sinus thrombosis (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Nerve root compression (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Peripheral nerve lesion (Nervous system disorders) | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Urethral haemorrhage (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Hypotension (Vascular disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panobinostat (N=129)
Anaemia (Blood and lymphatic system disorders) | 52
Leukopenia (Blood and lymphatic system disorders) | 16
Lymphopenia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 36
Thrombocytopenia (Blood and lymphatic system disorders) | 109
Bradycardia (Cardiac disorders) | 4
Palpitations (Cardiac disorders) | 4
Sinus tachycardia (Cardiac disorders) | 7
Tachycardia (Cardiac disorders) | 8
Hypothyroidism (Endocrine disorders) | 20
Abdominal distension (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 17
Abdominal pain lower (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 21
Aphthous stomatitis (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 25
Diarrhoea (Gastrointestinal disorders) | 96
Dry mouth (Gastrointestinal disorders) | 14
Dyspepsia (Gastrointestinal disorders) | 12
Flatulence (Gastrointestinal disorders) | 6
Gastritis (Gastrointestinal disorders) | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Gingival bleeding (Gastrointestinal disorders) | 5
Haemorrhoids (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 87
Stomatitis (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 55
Asthenia (General disorders) | 24
Chills (General disorders) | 8
Fatigue (General disorders) | 60
Influenza like illness (General disorders) | 4
Local swelling (General disorders) | 4
Non-cardiac chest pain (General disorders) | 10
Oedema peripheral (General disorders) | 17
Pyrexia (General disorders) | 56
Thirst (General disorders) | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 5
Bronchitis (Infections and infestations) | 4
Bronchopneumonia (Infections and infestations) | 6
Cystitis (Infections and infestations) | 3
Device related infection (Infections and infestations) | 3
Ear infection (Infections and infestations) | 3
Folliculitis (Infections and infestations) | 4
Herpes zoster (Infections and infestations) | 3
Influenza (Infections and infestations) | 8
Lower respiratory tract infection (Infections and infestations) | 7
Lung infection (Infections and infestations) | 5
Nail infection (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 12
Oral candidiasis (Infections and infestations) | 3
Oral herpes (Infections and infestations) | 5
Pneumonia (Infections and infestations) | 5
Respiratory tract infection (Infections and infestations) | 5
Rhinitis (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 9
Upper respiratory tract infection (Infections and infestations) | 19
Urinary tract infection (Infections and infestations) | 7
Contusion (Injury, poisoning and procedural complications) | 7
Alanine aminotransferase increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 6
Blood alkaline phosphatase increased (Investigations) | 7
Blood creatine phosphokinase increased (Investigations) | 3
Blood creatinine increased (Investigations) | 10
Blood potassium decreased (Investigations) | 4
Blood thyroid stimulating hormone increased (Investigations) | 3
Electrocardiogram QT prolonged (Investigations) | 4
Electrocardiogram T wave inversion (Investigations) | 3
Gamma-glutamyltransferase increased (Investigations) | 4
Platelet count decreased (Investigations) | 4
Weight decreased (Investigations) | 16
Decreased appetite (Metabolism and nutrition disorders) | 48
Dehydration (Metabolism and nutrition disorders) | 7
Fluid retention (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 19
Hypomagnesaemia (Metabolism and nutrition disorders) | 7
Hyponatraemia (Metabolism and nutrition disorders) | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 24
Bone pain (Musculoskeletal and connective tissue disorders) | 10
Muscle spasms (Musculoskeletal and connective tissue disorders) | 30
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 13
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Dizziness (Nervous system disorders) | 8
Dysgeusia (Nervous system disorders) | 21
Headache (Nervous system disorders) | 27
Lethargy (Nervous system disorders) | 9
Neuralgia (Nervous system disorders) | 5
Paraesthesia (Nervous system disorders) | 3
Sinus headache (Nervous system disorders) | 4
Somnolence (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 5
Anxiety (Psychiatric disorders) | 16
Confusional state (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 11
Insomnia (Psychiatric disorders) | 12
Dysuria (Renal and urinary disorders) | 5
Haematuria (Renal and urinary disorders) | 4
Vaginal haemorrhage (Reproductive system and breast disorders) | 4
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 36
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 10
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 8
Dry skin (Skin and subcutaneous tissue disorders) | 13
Erythema (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Night sweats (Skin and subcutaneous tissue disorders) | 4
Petechiae (Skin and subcutaneous tissue disorders) | 12
Pruritus (Skin and subcutaneous tissue disorders) | 21
Rash (Skin and subcutaneous tissue disorders) | 11
Haematoma (Vascular disorders) | 5
Hypotension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.